CLINICAL TRIAL: NCT04891094
Title: Lung and Diaphragm Ultrasound in the Early Postoperative Course Following Lung Transplantation
Acronym: LUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Michael Zoller MD, Clinical Professor, Ludwig-Maximilians - University of Munich
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LMU 283-16
Record Dates: First submitted 2021-02-18; First posted 2021-05-18 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Lung Transplantation
Keywords: Lung ultrasound; Lung transplantation; primary graft dysfunction; Lung Sliding
MeSH Terms: conditions — Primary Graft Dysfunction | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ultrasound — daily ultrasound of the lung and the diaphragm

SUMMARY:
This feasibility study tries to define the value of daily Lung and Diaphragm Ultrasound in the early postoperative course following Lung transplantation by comparing its diagnostic accuracy with that of standard of care diagnostic procedures

DETAILED DESCRIPTION:
Lung transplantation remains a high risk procedure. Common complications in the early postoperative course are, among others, primary graft dysfunction (PGD), hemorrhage, anastomosis insufficiency leading to pneumothorax, pneumonia, atelectasis and diaphragm dysfunction. Early diagnosis of complications is important to avoid further deterioration. Lung ultrasound (LUS) and diaphragm ultrasound (DUS) has a high diagnostic accuracy for identifying frequent conditions in the critically ill. Studies evaluating its value in patients following lung transplantation are missing. This study investigates the feasibility and clinical ability of LUS and DUS to identify common complications following lung transplantation and compares it to standard of care diagnostic procedures. The investigators start a prospective cohort study of lung transplant recipients who undergo lung transplantation at the university hospital Munich. Daily LUS and DUS in the early postoperative phase will be performed to detect and monitor complications. The US results will be compared to the results of diagnostic procedures of the clinical routine such as clinical examination, chest x ray, hemodynamic monitoring, expert opinion on PGD and laboratory parameters.

The hypothesis is that daily LUS and DUS following lung transplantation helps to diagnose complications early and with higher accuracy compared to the results of diagnostic procedures of the clinical routine.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* patient following lung transplantation

Exclusion Criteria:

* no informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-04-16 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
The value of LUS in diagnosing PGD | postoperative day 3
  number of days with PGD in LUS versus standard of care
Is Lung Sliding reliable in the early postoperative course following lung transplantation? | postoperative day 3
  Number of days with detectable lung sliding in LUS. Number of days with detectable pneumothorax in LUS.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anaesthesiology of the University Hospital of Munich, Munich, Germany

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR